CLINICAL TRIAL: NCT04259047
Title: Health Beliefs, Glycemic Control, and Preventing Cognitive Decline in African Americans with Diabetes and Mild Cognitive Impairment: a Randomized Clinical Trial
Acronym: DREAM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Barry Rovner, Principal Investigator, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01AG065467 (NIH)
Record Dates: First submitted 2020-02-05; First posted 2020-02-06 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Mild Cognitive Impairment; Diabetes
Keywords: Mild Cognitive Impairment; Diabetes; African American; Health Disparities; Retinal Imaging
MeSH Terms: conditions — Cognitive Dysfunction; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: This RCT will be double-masked in that all participants will receive an active intervention, and investigators and outcome assessors will be masked to treatment assignment. To maintain masking: 1) the Outcome Assessor will be masked to treatment assignment; 2) interventionists who deliver study treatments gather no outcome data; and 3) only primary care physicians (PCPs) who treat participants in the active group[, and the Study Coordinator, Project Director, and Statistician will be unmasked. Because the 2 interventions (DREAM and EUC) share identifying characteristics (i.e., in-home delivery by CHWs, same educational materials, same visit frequency), the risk of unmasking is reduced. At each outcome assessment, the Outcome Assessor will instruct participants on the purpose and importance of maintaining masking, and will request that they reveal no information about their study participation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diabetes Regulation for Eyesight and Memory (DREAM) (Experimental): DREAM is a behavioral treatment for diabetes mellitus (DM), as well as a secondary prevention strategy for dementia. DREAM acts to reinforce DM self-care and address negative beliefs about medications and physicians, which compromise glycemic control in African Americans (AAs). In DREAM, race-concordant community health workers (CHWs) will: 1) deliver in-home DM education tailored to AAs with MCI; 2) use action plans to reinforce diabetes self-care; 3) facilitate telehealth visits with a DM nurse educator to improve DM self-care and address participants' health beliefs; and 4) increase primary care physicians' (PCP) awareness of participants' cognitive deficits and health beliefs to optimize treatment of DM. .
  Interventions: Behavioral: Diabetes Regulation for Eyesight and Memory
- Enhanced Usual Care (EUC) (Active Comparator): EUC consists of home visits by a CHW in which general DM education is provided.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Diabetes Regulation for Eyesight and Memory — Participants randomized to DREAM will have 11 in-home visits over 2 years with a CHW, and 4 telehealth visits with a DM nurse educator.
  Other Names: DREAM
  Arms: Diabetes Regulation for Eyesight and Memory (DREAM)
Behavioral: Enhanced Usual Care — Participants in this group will have 11 in-home CHW visits over 24 months to control for attention. During these visits, the CHW will provide general diabetes education. There will be no telehealth visits.
  Other Names: EUC
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
This double-masked, 2-year, single-site, phase II RCT will test the efficacy of DREAM (Diabetes Regulation for Eye Sight and Memory to prevent cognitive decline in African Americans (AAs) with amnestic multiple domain mild cognitive impairment (MCI) and poorly controlled diabetes (i.e., hemoglobin A1c [HbA1c] level ≥ 7.5%). Participants will be randomized to DREAM [11 home-based treatment sessions with a community health worker (CHW), and 4 telehealth visits with a Diabetes Nurse Educator over 2 years] or Enhanced Usual Care (EUC), which is usual care enhanced with home-based diabetes education. The primary outcome is decline in verbal memory over 2 years. Follow-up data will be collected at 6, 12, 18, and 24 months. In addition, participants will have ophthalmology assessments (at Wills) at baseline, 12 and 24 months to determine whether retinal Vessel Area Density, and/or Retinal Nerve Fiber Layer thickness mediate DREAM's treatment effect.

DETAILED DESCRIPTION:
Thirty percent of African Americans (AAs) with Mild Cognitive Impairment (MCI) have (DM), which increases risk for cognitive decline and dementia. Poorly controlled DM magnifies this risk, and AAs have worse glycemic control than Whites. This single-site, double-blind, active-control, phase II randomized controlled trial (RCT) will compare the efficacy of DM-Specific Behavioral Activation (DM-BA) vs. Enhanced Usual Care (EUC) to prevent decline in verbal memory (primary outcome) over 2 years in 200 AAs over age 65 years with amnestic multiple-domain MCI and poorly controlled DM. DM-BA is a behavioral treatment for DM, as well as a secondary prevention strategy for dementia. DM-BA reinforces DM self-care and addresses negative beliefs about medications and physicians. In DM-BA, race-concordant community health workers (CHWs) will: 1) deliver in-home DM education tailored to AAs with MCI; 2) use action plans to reinforce DM self-care; 3) facilitate telehealth visits with a DM nurse educator to guide management of DM and address participants' health beliefs; and 4) increase primary care physicians' (PCP) awareness of participants' cognitive deficits and health beliefs to optimize treatment of DM. The control treatment, EUC, is usual medical care enhanced with DM self-care education. Both DM-BA and EUC deliver DM education and have the same number of in-home treatment visits (i.e., 6 visits over 6 months, and 5 booster visits over the next 18 months). EUC, however, does not include DM-BA's behavioral approach to improve glycemic control, telehealth visits with a DM nurse educator, or PCP communication. The treatment comparison will identify DM-BA's specific efficacy over and above EUC. Randomization will follow a fixed scheme with a 1:1 allocation ratio and stratification by hemoglobin A1c level (7.5% - 9% vs. ≥ 9%). We are recruiting participants from primary care practices. We will administer the Hopkins Verbal Learning Test-Revised (HVLT-R) (to assess verbal memory; the primary outcome) and the Uniform Data Set neuropsychological battery (to assess executive function, processing speed, language, visuospatial function, and global cognition; all exploratory outcomes) at baseline and months 6, 12, 18, and 24. The primary efficacy analysis will compare trajectories in HVLT-R Total Recall scores over 2 years by treatment group. A novel exploratory aim will investigate whether Optical Coherence Tomography (OCT) measures of retinal Vessel Area Density (an indicator of microvascular disease) and/or Retinal Nerve Fiber Layer thickness (an indicator of neurodegeneration) [i.e., proxies for cerebral microvascular and neurodegenerative disease, respectively] mediate treatment effects. We will also explore whether APOE genotype moderates treatment effects, and explore DM-BA's impact on multiple cognitive domains and incidence rates of dementia. We powered this RCT to test the hypothesis that the slope of the trajectory of HVLT-R Total Recall scores in DM-BA participants will not differ significantly from 0 (i.e., no change), whereas the slope of the trajectory of HVLT-R Total Recall scores in EUC controls will be significantly negative (i.e., decline) over 2 years. With 25% attrition over 2 years, a randomized sample of 200 participants will provide over 80% power for detecting an annual 1-point difference in slopes (2-point difference in 2-year means; a clinically meaningful difference) at the two-sided alpha=0.05 level. The scientific rigor of this study derives from the double-blind RCT design; recruitment of a sample at high risk for cognitive decline; use of validated outcome measures; adequate power; masked outcome assessments; delivery of two standardized credible interventions, and data already demonstrating DM-BA's effectiveness to improve glycemic control. This RCT is innovative because it will determine whether improving glycemic control prevents cognitive decline in a high risk population. Previous RCTs have studied lower risk populations and have been inconclusive. We will also uniquely explore whether OCT-evidence of retinal microvascular disease and/or neurodegeneration mediate treatment effects. This RCT is significant because it targets two prevalent problems in older AAs with DM (i.e., poor glycemic control and dementia). AAs' high risk for this comorbidity emerges in part from cultural factors (e.g., health beliefs) and requires culturally relevant treatment. The number of older AAs with DM in the U.S. (now 1 million) will double by 2030. This doubling will increase the burden of dementia in AAs (who already have twice the rate of dementia as Whites) and necessitates preventive treatment. We have the experience and expertise to test this treatment, and the opportunity to change how DM is treated to prevent cognitive decline in AAs with DM. If successful, this RCT will bring us closer to achieving health equity for all Americans and meet the goals of the National Alzheimer's Project Act.

ELIGIBILITY:
Inclusion Criteria:

* African American race
* Age ≥ 65 years
* Type 2 DM
* Duration of DM ≥ 1 year
* HbA1c ≥ 7.5
* Amnestic multiple-domain MCI by NIA-AA criteria
* Able to provide written informed consent

Exclusion Criteria:

* Dementia
* Excluded medical conditions
* Life expectancy less than two years in the opinion of the PCP
* Psychiatric disorders
* Cannot provide written consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 145 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Decline in Verbal Memory | 24 months
  Scores on the Hopkins Verbal Learning Test total recall (HVLT)

OTHER OUTCOMES:
Glycemic Control | 24 months
  Hemoglobin A1c (HbA1c)
Retinal Vessel Area Density Layer thickness mediates treatment effects; | 24 months
  Retinal Vessel Area Density
Retinal Nerve Fiber Layer Thickness Layer thickness mediates treatment effects; | 24 months
  Retinal Nerve Fiber Layer Thickness
Dementia | 24 months
  Incidence of dementia based on an adjudication panel

CONTACTS AND LOCATIONS:
Overall Officials: Barry Rovner, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Casten R, Leiby BE, Kelley M, Rovner BW. A randomized controlled trial to test the efficacy of a diabetes behavioral intervention to prevent memory decline in older blacks/African Americans with diabetes and mild cognitive impairment. Contemp Clin Trials. 2022 Dec;123:106977. doi: 10.1016/j.cct.2022.106977. Epub 2022 Oct 28. PMID 36341847